CLINICAL TRIAL: NCT02892097
Title: Examining the Effects of Transcranial Direct Current Stimulation and Task-specific Practice on Cortical Modulation Among Individuals With Unilateral Spatial Neglect Post Stroke
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Task-Specific Practice for Post-stroke Neglect
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrolled 1 participant, PI left the institution.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00056688; P2CHD086844 (NIH)
Record Dates: First submitted 2016-08-10; First posted 2016-09-08 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Hemispatial Neglect
Keywords: tDCS; neglect; paresis; transcranial direct current stimulation; rehabilitation
MeSH Terms: conditions — Stroke; Perceptual Disorders; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parietal tDCS plus RTP (Active Comparator): Single session of bilateral parietal tDCS (2.0 mA for 30 minutes) paired with repetitive task-specific practice (RTP).
  Interventions: Device: tDCS; Behavioral: Repetitive task-specific practice (RTP)
- Primary motor cortex tDCS plus RTP (Active Comparator): Single session of bilateral primary motor cortex tDCS (2.0 mA for 30 minutes) paired with repetitive task-specific practice (RTP)
  Interventions: Device: tDCS; Behavioral: Repetitive task-specific practice (RTP)
- Sham tDCS plus RTP (Sham Comparator): Single session of sham tDCS (for 30 minutes) paired with repetitive task-specific practice (RTP)
  Interventions: Device: sham tDCS; Behavioral: Repetitive task-specific practice (RTP)

INTERVENTIONS:
Device: tDCS — tDCS is a form of noninvasive brain stimulation. Electrodes are placed on the scalp (parietal or primary motor cortex) and deliver a low level of direct current (2mA). tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand.
  Other Names: noninvasive brain stimulation; transcranial direct current stimulation
  Arms: Parietal tDCS plus RTP; Primary motor cortex tDCS plus RTP
Device: sham tDCS — Sham tDCS will be delivered for 30 minutes in conjunction with repetitive task-specific practice for the arm/hand.
  Arms: Sham tDCS plus RTP
Behavioral: Repetitive task-specific practice (RTP) — Participants will practice using their paretic arm/hand to complete functional movements during each (3) 30 minute training session.
  Other Names: task practice

SUMMARY:
The purpose of this study is to test the effects of three different rehabilitation training sessions that combine non-invasive brain stimulation (transcranial direct current stimulation, tDCS) with arm rehabilitation training (repetitive task-specific practice, RTP) for individuals with unilateral spatial neglect following stroke. This study is designed to determine the effects of tDCS + RTP on the excitability in the brain, attention to the affected side, and arm movement ability.

DETAILED DESCRIPTION:
Unilateral neglect (neglect) is common after stroke and is characterized by an inattention to one side of the body or environment. There is growing evidence that disconnections to fronto-parietal neural networks in the lesioned hemisphere not only cause neglect, but also cause these same networks to be hyperexcited in the non-lesioned hemisphere. Individuals with neglect typically experience motor impairments also since the regions of the brain that control attention also control movement.

Transcranial direct current stimulation (tDCS) when paired with repetitive task-specific practice (RTP) has the potential to modulate cortical activity (fronto-parietal networks) and facilitate motor and attentional recovery for individuals with neglect since tDCS can modulate the excitability of targeted cortical regions. tDCS is a form on non-invasive brain stimulation and RTP is the gold standard post-stroke motor recovery intervention.

It is particularly important investigators examine the effect of RTP + tDCS on cortical modulation in order to understand the underlying mechanism of the intervention and determine whether RTP+ tDCS (parietal or primary motor cortex [M1]) promotes greater neural modulation than RTP alone. Traditionally, electrodes are placed on M1 to facilitate motor recovery and on the parietal lobe to facilitate attentional recovery, however this intervention is designed to target each of these impairments (motor, attention) and enhance cortical modulation of fronto-parietal networks. Therefore, investigators must also determine the optimal electrode montage and placement for pairing tDCS with RTP for individuals with neglect.

The purpose of the proposed pilot project is to examine the effects of transcranial direct current stimulation (tDCS) paired with repetitive task-specific practice (RTP) on modulation of fronto-parietal network connectivity (measured by transcranial magnetic stimulation [TMS]), motor impairment (measured with kinematic assessment), and attentional impairment (measured with Behavioral Inattention Test) among individuals with unilateral neglect and hemiparesis post stroke. This three day cross-over design study will examine the optimal electrode placement and montage using 3 conditions: (1) tDCS to parietal lobe + RTP (2) tDCS to primary motor cortex + RTP (3) sham tDCS + RTP.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hemispheric ischemic stroke or hemorrhagic subcortical stroke ≥3 months post stroke (lesion type and location to be confirmed with MRI)
* Neglect (Virtual Reality Lateralized Attention Test score <18)
* Upper extremity Fugl-Meyer score between 20-56/60
* Inducible motor evoked potential (MEP) of the abductor pollicis brevis (APB) on the affected side using transcranial magnetic stimulation (TMS)
* ≥18 years old

Exclusion Criteria:

* History of cortical hemorrhagic stroke
* Severe spasticity (Modified Ashworth Scale score ≥3) in paretic upper extremity
* Severe aphasia limiting participant's ability to follow 2 step directions
* History of seizures
* History of brain tumor
* History of skull defect
* Hardware in skull or spine (e.g. coils, clips)
* Implantable medical device (e.g. pacemaker)
* Metal in body that is not compatible with MRI
* Pregnant (women of child bearing age will be asked if they are pregnant or could possibly be pregnant)
* Unable to travel to Upper Extremity Motor Function Laboratory at the Center for Rehabilitation Research in Neurological Conditions
* Currently enrolled in another study using transcranial direct current stimulation (tDCS) or transcranial magnetic stimulation (TMS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Change in excitability of fronto-parietal connectivity | Participants will be assessed at baseline and 30 minutes later (immediately following intervention session).
  Excitability of fronto-parietal connectivity measured by paired pulse twin coil transcranial magnetic stimulation (TMS) test. In each session, the difference in excitability of fronto-parietal connectivity between pre and post stimulation will be measured.

SECONDARY OUTCOMES:
Change in kinematics | Participants will be assessed at baseline and 1 hour later (immediately following intervention session).
  A kinematic assessment will be conducted to assess changes in motor impairment.
Change on Behavioral Inattention Test | Participants will be assessed at baseline and 1.5 hours later (immediately following intervention session).
  A neglect assessment will be conducted to assess changes in attentional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Grattan, PhD, OTR/L, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No